CLINICAL TRIAL: NCT05330221
Title: ACHIEVE GREATER: Addressing Cardiometabolic Health In Populations Through Early PreVEntion in the GREAT LakEs Region
Brief Title: Project 2: ACHIEVE- HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, David Lanfear, Section Head - Advanced Heart Failure and Transplant Cardiology, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WSU22115
Record Dates: First submitted 2022-03-21; First posted 2022-04-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Hypertension
Keywords: Prevention; Heart Failure
MeSH Terms: conditions — Heart Failure; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): PAL2 Intervention
  Drug Therapy
  Interventions: Behavioral: PAL2; Drug: PHARM-PAL2
- Usual Care Group (No Intervention): Participants that are randomized into usual care will be assisted with arrangement of follow-up, either with existing primary care provider (PCP) or a Wayne Health provider. All subsequent medical treatment will be at the discretion of the PCP.

INTERVENTIONS:
Behavioral: PAL2 — Community health worked based intervention to mitigate psychosocial and life circumstance barriers to optimize health promotion coupled with high blood pressure and lifestyle disease state education Other Names: Pragmatic personalized, adaptable approach to lifestyle and life circumstance
  Arms: Intervention Group
Drug: PHARM-PAL2 — All intervention arm participants will be referred to our study pharmacist who will prescribe a antihypertensive medication as per standard of care medical treatment algorithm to achieve BP control.
  Per AHA recommended guidelines, participants with an indication of diabetes mellitus (DM) and/or CKD will be started on SGLT2 inhibitor within the first month of starting the study intervention.
  Arms: Intervention Group

SUMMARY:
This project is part of the ACHIEVE GREATER (Addressing Cardiometabolic Health In Populations Through Early PreVEntion in the GREAT LakEs Region) Center (IRB 100221MP2A), the purpose of which is to reduce cardiometabolic health disparities in two cities: Detroit, Michigan, and Cleveland, Ohio. The ACHIEVE GREATER Center involves four separate but related projects that aim to mitigate health disparities in risk factor control for three chronic conditions, hypertension (HTN, Project 1), heart failure (HF, Projects 2 and 4) and coronary heart disease (CHD, Project 3). The first three projects will involve the use of Community Health Workers (CHWs) to deliver an evidence-based practice intervention program called PAL2. Projects 1-3 also utilize the PAL2 Implementation Intervention (PAL2-II), which is a set of structured training and evaluation strategies designed to optimize CHW competence and adherence (i.e., fidelity) to the PAL2 intervention program. The present study is Project 2 of the ACHIEVE GREATER Center.

DETAILED DESCRIPTION:
Heart failure (HF) is one of the most common, costly, and deadly diseases affecting humans. Hypertension is the largest single risk factor for HF, accounting for over half of all new cases. Accordingly, early interventions to prevent HF, in particular blood pressure (BP) control, are critical. However, implementation of effective treatments remains suboptimal, especially in Detroit, Michigan. To better engage the at-risk community, the team developed an innovative mobile health unit (MHU) program that uses geospatial health and area-level exposure data to direct health services to communities in highest need, who may not otherwise engage with traditional health care settings. Another key to preventing HF is usage of guideline-directed medical therapy (GDMT), not only for treating high BP, but also providing medications proven to reduce HF incidence. In particular, inhibitors of sodium-glucose transporter type 2 (SGLT2) prevent HF and loss of kidney function in at-risk patients. Yet, these are dramatically under-utilized, further contributing to health disparities. Project 2 of ACHIEVE GREATER uses a pragmatic, randomized, unblinded, clinical trial to implement and test a novel intervention leveraging our MHU platform to improve care access combined with enhanced collaborative care delivery among patients with Stage A HF (defined as asymptomatic individuals with known pre-conditions such as hypertension who are at-risk for later-stage clinical HF). The key components of the program are 1) a personalized intervention conducted by community health workers that links patients with available community resources, and 2) pharmacist-directed therapy optimization per a standardized GDMT protocol. This intervention will address multiple domains and levels of impact to reduce the large gaps in care of stage-A HF patients in the community and prevent progression towards symptomatic HF.

ELIGIBILITY:
Inclusion:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Detroit-area resident (defined as those who attended a Detroit-area community event)
2. ≥18 years of age
3. At least one of the following:

A) Screening systolic BP ≥ 140 and/or diastolic BP ≥ 90 mm Hg OR

B) Screening BP 130-139 mm Hg plus ≥1 additional HF risk factors:

i. Diabetes (HbA1c ≥ 6.5%) ii. CKD stage 3(i.e. eGFR 30-60 mL/min/m2) OR C) Treated (1-2 antihypertensive medications) stage 1 HTN (systolic BP 130-139 and/or diastolic BP 80-89) with or without >1 additional HF risk factors OR

D) Treated stage 1 HTN w/ systolic BP 120-129 with additional HF risk factors:

i. Diabetes (HbA1c ≥ 6.5%) ii. CKD stage 3(i.e. eGFR 30-60 mL/min/m2)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Previous diagnosis of HF
2. Uncontrolled diabetes (HbA1C ≥8.0% from SOC screening labs)
3. Chronic use of insulin or >1 anti-diabetic medication
4. Self-reported pregnancy (or planning to become pregnant in the next year)
5. Severely uncontrolled BP at screening visits (SBP ≥180 mm Hg and/or diastolic BP ≥110 mmHg)
6. Point of care (POC) BNP measurement ≥400 ng/L. If POC BNP was not obtained, then NTproBNP ≥ 1000 ng/L from screening labs will be excluded.
7. eGFR <45 ml/min/sq-m on SOC screening labs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (BP) | 12 months
  Change in systolic BP at 12-months vs. baseline (detect ≥ 5 mm Hg difference). This will be determined by comparing the "post-trial systolic BP" at 12-month mobile health unit (MHU) visit versus the "baseline systolic BP" at screening MHU visit.
NT-proB-type Natriuretic Peptide (NT-proBNP) | 12 months
  Change in NT-proBNP over 12 months

SECONDARY OUTCOMES:
Utilization rates for anti-RAS medications and SGLT2 inhibitors | 12 months
  Utilization rates for anti-RAS medications (ACE-inhibitors, angiotensin receptor blockers, ARNi's) and SGLT2 inhibitors in the intervention group compared to usual care at the 12-month visit.
Geospatial outreach | 24 months
  Reach will be assessed by evaluating the number of patients who are screened by the MHUs; the number and percentage of screened patients who meet inclusion and exclusion criteria for ACHIEVE- HF; the number and percentage of patients who meet inclusion that enroll; and the number and percentage of enrolled patients who do and do not complete the study. For each of these measures, qualitative and quantitative methods will be utilized to understand how patient and community level characteristics may have contributed to higher or lower indicators of reach.

OTHER OUTCOMES:
Patient satisfaction | 24 months
  Patient satisfaction will be evaluated by questionnaires administered at months 12 and 24.
Patient wellbeing | 24 months
  The impact of the Pharm-PAL2 intervention on quality of life and wellbeing will be evaluated by questionnaires administered at months 12 and 24.
Cost effectiveness | 12 months
  Cost Effectiveness of the Pharm-PAL2 intervention will determined using disaggregated cost analysis, assessing the cost of intermediate inputs per endpoint achieved with BP and NT-proBNP evaluated separately, providing a detailed breakdown of resources used. To allow some cross-intervention benchmarking, the investigators additionally estimate the cost per quality adjusted life years (QALY) extended by the intervention
The number of hospitalizations, emergency department visits and deaths | 12 months
  To evaluate the effectiveness of the Pharm-PAL2 intervention to reduce CVD related hospitalizations, emergency department visits and death.
BP Control (<130/80) | 12 months
  To determine the proportion of participants with controlled BP (<130/80) at the 12 month visit.
NT pro BNP (> 125 ng/L) | 12 months
  To determine the proportion of participants with elevated NT pro BNP (> 125ng/L) at the 12 month visit.
Change in creatinine | 12 months
  To determine the effectiveness of the Pharm-PAL2 intervention to improve kidney function (measured by change in creatinine) at the 12-month visit compared to baseline.
Change in glycated hemoglobin | 12 months
  To determine the effectiveness of the Pharm-PAL2 intervention to improve diabetes control (measured by change in glycated hemoglobin) at the 12-month visit compared to baseline.
Utilization rates of other cardiovascular medications | 24 months
  To examine the effectiveness of the Pharm-PAL2 intervention to improve utilization rates of other cardiovascular medications of interest (e.g. statins, measured by the rate of prescription of statins).

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States